CLINICAL TRIAL: NCT02549066
Title: Impact of CArdiopulmonary Bypass Flow on Renal Blood Flow, Function and OXygenation
Acronym: ICAROX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lukas Lannemyr, M D, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SahlgrenskaUHThoraxLL4
Record Dates: First submitted 2015-09-11; First posted 2015-09-14 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Complication of Extracorporeal Circulation; Kidney Circulation Disorder; Renal Function Disorder
Keywords: cardiopulmonary bypass; renal blood flow; renal function; renal oxygenation
MeSH Terms: interventions — Milrinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Increased cardiopulmonary bypass flow — In randomized order, CPB flow will be adjusted to 2,4, 2,7 and 3,0 L/min/m2. After 10 minutes of steady conditions at each level, measurements will be made.
Drug: Milrinone — After weaning from CPB, patients with signs of cardiac failure (as defined below) will be given milrinone (0,04 mg/kg as a loading dose and 0,50 ug/kg/min as subsequent infusion). Measurements of systemic and renal variables will be made before and 30 minutes after the dose.
  Indication: Central venous pressure (CVP) ≥ 12 mmHg AND/OR Pulmonary Capillary Wedge Pressure (PCWP) ≥ 16 mmHg AND Cardiac Index (CI) ≤ 2,1 L/min/m2 AND Pulse Pressure Variation (PPV) < 12 %.
  Other Names: Inotrope

SUMMARY:
Cardiac surgery with cardiopulmonary bypass (CPB), especially when oxygen delivery is low, is associated with acute kidney injury. Unpublished data shows that renal oxygen delivery is compromised during CPB due to low hematocrit and redistribution of blood flow away from the kidneys. We wish to study if increased CPB flow can improve renal oxygenation.

Patients who develop cardiac failure after weaning from CPB will be treated as per our departments routine with the inotropic agent milrinone, and measurements will be made before and after treatment.

DETAILED DESCRIPTION:
Acute kidney injury (AKI), defined as a 50 % increase in serum creatinine above baseline, is a complication commonly seen in the intensive care unit. After cardiac surgery with cardiopulmonary bypass, up to 30% of the patients develop AKI and about 2-5% requires acute dialysis. AKI renders increased morbidity, mortality and costs, and the mortality rate increases with the degree of renal impairment.

The development of AKI is considered to be a multifactorial process, where renal ischemia, nephrotoxic agents and inflammatory processes all contribute. Oxygen delivery to the kidney is compromised in states of low cardiac output, severe hypotension and anemia. The renal medulla, utilizing large amounts of oxygen in the tubular sodium reabsorption mechanism, is hypoxic already under normal conditions and therefore especially susceptible to acute renal ischemia. In postoperative AKI, Redfors et al showed that renal vasoconstriction in combination with high medullary oxygen consumption deteriorates the oxygen supply-demand relationship. This supply-demand mismatch of the renal oxygenation is considered a key mechanism of medullary ischemia.

The use of cardiopulmonary bypass (CPB) in cardiac surgery is associated with AKI, but the mechanisms remain unclear. Institution of CPB changes vasomotor tone and decreases renal perfusion pressure. Hemodilution during CPB could potentially improve microcirculatory flow through reduced blood viscosity, but it might also reduce the oxygen delivery to the renal medulla. The extracorporeal circulation triggers the systemic inflammatory response syndrome, contribute to hemolysis and micro embolization, all with negative renal effects.

de Somer and co-workers recently showed that during CPB, a nadir delivery of oxygen (DO2) of < 262 mL/minute/m2 is independently associated with AKI. This emphasizes the importance of oxygen delivery. Preliminary data from a recent study indicates that CPB induces a significant renal oxygen demand/supply mismatch due to a 25% fall in renal oxygen delivery (RDO2), in turn caused by a haemodilution and redistribution of RBF away from the kidneys.

CPB flow-rates varies between different centres depending mainly on empirical experience. Common flow-rates at the institution of CPB; 2,2-2,5 L/minute/m2 equals the average cardiac index in anesthetized adults with normal hematocrit. Potential benefit from low flow is less oedema, less haemolysis, less hypertension during hypothermic CPB and reduction of the bronchial blood flow that rewarms the heart and might obscure the surgeons view. Increased CPB flow is routinely used when indications of inadequate perfusion such as lactataemia, increased pCO2 or low central venous oxygen saturation (SvO2) is seen. Mackay and co-workers showed that increased CPB flow significantly increased renal perfusion during normothermic CPB in pigs. Adluri et al found that higher pump flow during hypothermic CPB in man increased hepatic blood flow. However, the impact of higher than usual flow rates on renal hemodynamics and oxygenation has not been studied in man.

We aim to study the impact of increased CPB flow on renal oxygenation, filtration fraction and blood flow. Renal vein and pulmonary artery catheters will be inserted after the start of anesthesia. During stable conditions after the start of CPB and aortic cross clamp, the CPB flow will be altered in a randomized fashion. Measurements will be made at three different CPB flows, ranging from our clinical standard 2,4 L/min/m2 up to 3,0 L/min/m2. Additional measurements will be made after weaning from CPB.

Cardiac failure requiring inotropic support after weaning from CPB is not uncommon. In our department, the drug of choice is milrinone. The effects of milrinone on systemic circulation has been well established, but the renal effects has not been studied in a clinical setting.

In patients requiring inotropic support after CPB using the criteria below milrinone will be administered (0,04 mg/kg as a loading dose and 0,50 ug/kg/min as subsequent infusion). Measurements of systemic and renal variables will be made before and 30 minutes after the dose.

Indication: Central venous pressure (CVP) ≥ 12 mmHg AND/OR Pulmonary Capillary Wedge Pressure (PCWP) ≥ 16 mmHg AND Cardiac Index (CI) ≤ 2,1 L/min/m2 AND Pulse Pressure Variation (PPV) < 12 %.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Scheduled cardiac surgery (Coronary Artery Bypass Grafting or Valve Replacement)
* Normothermia during cardiopulmonary bypass
* Normal preoperative serum creatinine (in men; 60-105 umol/L, in women 45-90 umol/L)

Exclusion Criteria:

* Left ventricular ejection fraction < 50%
* Body mass index > 32 kg/m2
* Previous cerebrovascular lesion
* Radiocontrast allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Renal oxygenation | 10 minutes
  Renal oxygen extraction measured as difference between arterial and renal vein blood oxygen content divided by arterial oxygen content.

SECONDARY OUTCOMES:
Renal oxygenation measured with Near InfraRed Spectroscopy (NIRS) | 10 minutes
  NIRS pads will be placed over the kidneys using ultrasound for guidance. Tissue oxygenation will be measured online during the whole study. NIRS measurements will be compared with renal oxygen extraction.
Filtration fraction | 10 minutes
  Renal extraction of 51-Cr-EDTA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of thoracic anesthesia, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lannemyr L, Bragadottir G, Redfors B, Ricksten SE. Effects of milrinone on renal perfusion, filtration and oxygenation in patients with acute heart failure and low cardiac output early after cardiac surgery. J Crit Care. 2020 Jun;57:225-230. doi: 10.1016/j.jcrc.2019.12.022. Epub 2020 Jan 6. PMID 31919012